CLINICAL TRIAL: NCT05985096
Title: The Effects of Virtual Reality Education on Balance, Depression, Anxiety and Stress Parameters in Healthy Young Individuals
Brief Title: The Effects of Virtual Reality Education on Balance, Depression, Anxiety and Stress Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, HALİL YILMAZ, Assistant professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-2325
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Anxiety; Depression; Stress; Balanced
Keywords: Depression; Stress; Anxiety; Virtual reality glasses
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Adequate physical activity not only reduces depression, but also prevents the neural dysfunction that can occur as a result of depression. However, the level of physical activity among young people is not sufficient. Based on this fact, we believe that it is necessary to use 3D virtual reality applications to increase physical activity levels and exercise motivation.
  The aim of our study is to investigate the effect of virtual reality training on balance, depression, anxiety and stress parameters in healthy young people.
  Interventions: Diagnostic Test: Virtual reality group
- Control Group (No Intervention): The control group will perform individual exercise. The physical activity will be monitored with video recordings.

INTERVENTIONS:
Diagnostic Test: Virtual reality group — Participants in this group will be expected to meet their physical activity levels using the Oculus Quest 2 VR Goggles platform with Racket, Climb, Acron, Skiing, Cycling games.
  Arms: Virtual Reality Group

SUMMARY:
If we examine the demographic data of the 2021 reports of the Turkish Statistical Institute (TUIK), we can see that the young population between the ages of 15 and 24 is 12,971,289 people, which is 15.3% of the total population. Considering the proportion of young population in our country, the evaluation of physical activity level has an important place, while the proportion of female university students who achieved sufficient physical activity level according to the scoring of the International Physical Activity Questionnaire (UFAA) was 8.5%, while the proportion of male students was 28.1% in previous studies (Arslan 2015). ).

We know from previous studies that achieving an adequate level of physical activity directly reduces the body mass index and indirectly reduces the cardiovascular risk associated with obesity (Swift 2018). Exercise reduces depression levels and the effects of depression. Although the neural mechanisms are not very clear, there are some predictions for physical exercise to reduce the level of depression (Gujral 2017). The hippocampus is an important cognitive and sensory centre, and it has been reported that hippocampal volume decreases by 5% in depressed individuals (Cole 2011). Hippocampal volume has been reported to increase rapidly with exercise (Bugg 2012).

The brain region most affected in major depressive disorder is the prefrontal cortex. After the prefrontal cortex is affected, symptoms such as negative affect and learned helplessness appear (Pizagalli 2021). Experimental studies in mice have shown that treadmill training creates new synaptic pathways in the prefrontal cortex and hippocampus (Mu 2022).

Another brain region affected by depression is the corpus striatum. Loss of corpus striatum volume is observed in patients with major depression (Zhang 2020). The volume of the corpus striatum modulates when physical exercise reaches a sufficient level. (Rotttensteiner 2015).

Adequate levels of physical activity not only reduce depression, but also prevent neural dysfunction that can occur as a result of depression. However, young people do not get enough exercise. Based on this fact, we believe that it is necessary to use 3D virtual reality applications to increase physical activity levels and exercise motivation.

The aim of our study is to investigate the effect of virtual reality training on balance, depression, anxiety and stress parameters in healthy young people.

DETAILED DESCRIPTION:
Our work will last 6 weeks and is planned as exercise for 1 hour a day, 2 days a week.

Group 1: The control group will do individual exercise. The monitoring of the physical exercises will be done with video recordings.

Physical exercises Stick exercises: Shoulder stick (wand) exercises aim to perform shoulder range of motion exercises by supporting the sore arm with a solid arm. Use the stick to make forward, side, backward, outward and inward movements as shown in the picture. Count to 5 at the end of each movement and return to the beginning (Puendgsuwan 2008).

Codman exercises: Step forward with one foot and lean forward on a stable surface such as a table. Release your arm using the weight: move it back and forth like a pendulum. c) Circle clockwise and counterclockwise (Cunningham 2020).

Squat exercises: With feet open at shoulder height, the person's back is against the wall and positioned 10 cm in front of the wall. The rolling pin on the shoulder is grasped with the hands. The person faces forward. The movement is performed by bending the hip and knee joints without disturbing the straightness of the back and without touching the wall. Then return to starting position, keeping the spine straight and extending the hip and knee joints. Perform 3 sets of 10 repetitions (Kubo 2019).

Tandem walking exercise: A straight line is drawn on the floor. From the person, 10 steps are taken to follow this straight line with the heel of the front foot to the tip of the back foot. 3 sets of eyes open and 3 sets of eyes closed (Cruz 2021).

Group 2: Virtual reality group. People in this group will be expected to meet their physical activity levels with Racket, Climb, Acron, Skiing, Cycling games using the Oculus Quest 2 VR goggles platform.

Virtual reality games Racket: Nx is a new type of game in VR that pushes the boundaries of what you can do with a racket and a ball. The game takes place inside a giant glass dome, the walls of which are lit up with targets that you have to destroy with the cannon. But this is no ordinary ball. If you hit it hard, it will crash into a wall, roll over, and bulldozers will crush everything in its path. Use the racket's hammer beam to retreat or aim the next hit exactly where you want it. Targets appear in waves and the aim is to destroy them all before you run out of energy. But targets aren't the only thing in the arena. That's why you need to hit quickly and accurately. But in this game, the aim is to teach you how to control the ball perfectly. It is an alternative to coordination exercises.

Climbing: The aim of this game is to simulate climbing. It can be used as an alternative to strengthening the upper limbs. From exploring mountain environments to scaling urban environments, the game is also designed to have the dual effect of feeling the excitement of climbing without ropes and experiencing the landscapes as you climb to new heights.

Acron: In this game, you take on the role of a large, ancient tree that is the sole guardian of golden acorns. In this simulation, he uses an arsenal of unique abilities across seven different maps to try and prevent golden acorns from being stolen. We plan to use this simulation as an alternative to lower extremity strengthening exercises.

Skiing: Start with your feet shoulder-width apart, arms at eye level and bent 90°. Then swing your arms down and back while squatting. Don't squat too deep and squeeze your core. Finally, swing your arms back to their original position while standing. Continue to squat and swing your arms vigorously. The aim of this simulation is to provide an alternative to squatting and wand exercises.

Cycling: How to play: Stand upright, keeping your core strong and engaged, and start 'cycling' with your arms. There are also two ways to do circular arm movements: with the arms at your sides, mostly as regular arm cycling moves, which will focus on the shoulders, chest and triceps muscles, or as boxing speedbag moves, with the forearms side by side at face level, which will focus on the forearms, triceps muscles and shoulder blades. The aim of this simulation is to provide an alternative to balance, stick and Codman exercises.

Questionnaires and tests to be used for evaluation Depression-Anxiety Stress Scale 21 (DASS 21): It is estimated that by 2020, depression, stress and anxiety-related disorders will be the second most common disease in the world. The prevalence of these disorders can also have a significant negative impact on countries' health expenditure, social harmony, business life and individuals. This scale will be used to measure the depression burden of students.

Motivation scale for participation in physical activity: This 16-question questionnaire assesses an individual's motivation to participate in physical activity. Questions 1-6 of the survey form the individual causes, 7-12 form the environmental causes and questions 13-16 form the dimension of irrationality. Questions 3,9,13,14,15,16 are reverse coded.

Repetitive joint position sense test: The test is scored during arm elevation positions that include 90° shoulder flexion and 90° shoulder abduction movements. For the shoulder flexion assessment, the individual is asked to stand facing the millimetre paper taped to the wall. The laser cursor is positioned 5 cm above the elbow joint so that wrist and elbow movements do not affect the measurements. The subject is asked to flex the shoulder joint to 90°. This shoulder movement is measured by the physiotherapist using a goniometer and the person is asked to maintain this position for 10 seconds with eyes open. The projection of the laser cursor is marked on millimetre paper. The 90° position is repeated 3 times with the eyes open and the person is asked to memorise this position. It is then returned to the starting position and the subject's eyes are closed. He is asked to repeat the same movement 3 times and the projection of the laser cursor is marked. For the abduction movement, the subject is asked to turn sideways towards the wall, with the head turned towards the wall, bringing the arm to 90° abduction and the angle is measured with a goniometer. The projections of the laser cursor are also marked. The starting point is assumed to be 0 and the projections of the points on the x and y axes are measured during the angle repetition. The deviation is calculated using the formula c=√x2+y2 (Düzgün 2011).

Star Balance Test: The Star Balance Test, originally called the Star Excursion Balance Test, is a reliable tool for measuring dynamic balance. Designed for the assessment of lower extremity injuries and disorders, it is also widely used to assess dynamic balance in sport. In addition, the Star Excursion Balance Test has been shown to have a high coefficient of internal reliability, but its coefficients of validity have not been investigated. The test is based on the ability to reach the farthest possible distance on the supporting leg with the free leg in 8 different directions and is a very high quality measure of dynamic balance performance in sport (Gribble 2013). Before starting the test, a dry and quiet environment that is not affected by changing weather conditions should be selected for the test. This is the most basic requirement for a valid and reliable test between repeated measurements.

Required Equipment

* A minimum of 2×2 meters of flat, dry and suitable Ground
* Test manager and scoring chart
* Flat adhesive tape (minimum 8 meters)
* Ruler or Metre Application: 4 strips cut to 2 metres are placed on the floor at an angle of 45 degrees. The subject should be barefoot if possible. Shoes affect the reliability of the test in repeated tests. The athlete waits in the centre of the star shape (the point where the lines intersect). If the right foot is chosen as the reach foot, the test direction is clockwise. For the left foot, the direction is counter-clockwise. The hands should be at the waist during the test and the position of the hands should not change during the test. If this is not the case, the athlete places the hands on the waist, repeats whichever line is left, and continues the test. The athlete reaches out as far as he can with his foot and lightly touches the strip with the tip of his toe. He then returns to the starting position (hands around his waist, feet in the air, on one leg). Then the other line is walked and a total of 8 lines are completed in this way. Each time, the examiner makes a mark with a pencil to measure the maximum point that the subject can touch at a later time. After the whole process has been repeated 3 times with the right foot, the left foot is switched and the process is repeated 3 times (Shaffer 2013). At the end of the test, the participant records the distances reached in the Cartex.

Nelson Hand Reaction Test: The Nelson hand reaction test can be measured using the ruler method. The subject is seated in a chair with the forearm and hand resting relaxed on the table. The tips of the thumb and forefinger are placed 8-10 cm from the table so that they are approximately parallel on the outside. The tips of the thumb and index finger should be horizontal to each other. The examiner holds the tip of the ruler between the thumb and index finger of the subject. The subject is instructed to look directly at the concentration zone (the black area between lines 0.120 and 0.30) and to catch the ruler when it is released. There are 20 trials, each starting after the 'ready' command. The result is read from the line at the top of the subject's thumb after the subject has caught the ruler. The lowest 5 and the highest 5 trials are discarded and the average of the remaining 10 trials is recorded as the result. The digits on the time scale represent thousandths of a second. The results are recorded as 5/1000 seconds (Musabaşoğlu 2008).

Mini Best Test: This test is used to evaluate the balance. The Mini Best (DDS) test has 14 parameters. Anticipatory postural control (standing up from sitting; toes up; standing on one leg), reactive postural control (compensatory corrective stepping forward; compensatory corrective stepping backward; compensatory corrective stepping sideways), sensory orientation (standing position (feet together); eyes open, hard surface; standing position (feet together): eyes closed, spongy surface; tilt - eyes closed), dynamic gait (change of walking speed; walking with horizontal head movements; turning while walking; stepping over an obstacle; double The task is evaluated with timed get up & walk tests [ 3 metres walking).

Scoring: The test consists of 14 items, each scored from 0 to 2 out of a maximum of 28. "0' indicates the lowest level of function and '2' indicates the highest level of function. If the person requires the use of an assistive device for any item, that item is scored one level lower. If the person requires physical assistance to perform the item, score that item as "0". For item 3 (standing on one leg) and item 6 (compensatory stepping - lateral), record the score of only one side (low score). For item 3 (standing on one leg) take the best time from 2 attempts (each side separately). For item 14 (time to stand up and walk with double duty), the score should be reduced by one level if the person's gait slows by more than 10% between double duty and non-double duty SCI.

Measurement Evaluation and Statistical Analysis

1. Sample size: Gpower 3.1. determined by power analysis using the programme. In the analysis (α=0.05, power (1-β) = 0.80, effect size= 0.8, and at least n=26 people should be included in the groups. It was set at n=30 in case of dropout.
2. Number and names of groups in the study: Group 1: Control group Group 2: Virtual reality grou
3. Properties to be measured: Depression, anxiety, stress parameters Balance Repetitive joint position sense Participation in physical activity Motivation Hand reaction
4. Statistical analysis: The data in the study are analysed using 5 parameters (skewness-curvature, Std/Mean, Q-Q plots, histogram and Shapiro-Wilk test). The parameters with a score higher than 3 and a sufficient number of data are considered to be normally distributed and are presented as Mean±Standard Deviation (MEAN±STD).The Independent Samples T-test is used to compare two independent groups and the Related Samples T-test is used to compare dependent groups. Pearson correlation is used for correlation analysis of parametric data. Parameters with a score of 3 or less in the normal distribution analysis are considered non-parametric, and the Mann-Whitney U test is used for comparisons between two independent groups, the Wilcoxon test is used for comparisons between dependent groups, and Spearman Rho's correlation analysis is used for correlation analysis. In the study, α=0.05 and p<α are considered significant. The IBM SPSS 28.00 package programme will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering
* Being between 18-25 years old

Exclusion Criteria:

* Having a musculoskeletal disease
* Having a systemic (cardiovascular, neurological) disease
* Not attending the training sessions more than once

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-06-05 (Estimated)

PRIMARY OUTCOMES:
Decrease in depression, anxiety stress parameters | 6 weeks
  The specified parameters are calculated using the DASS 21 scale before and after the intervention.

SECONDARY OUTCOMES:
Increased hand reaction | 6 weeks
  Before and after the intervention, specified parameters are measured using the Nelson Hand Reaction Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University Faculty of Medicine Department of Anatomy, Ordu, Black Sea, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bugg JM, Shah K, Villareal DT, Head D. Cognitive and neural correlates of aerobic fitness in obese older adults. Exp Aging Res. 2012;38(2):131-45. doi: 10.1080/0361073X.2012.659995. PMID 22404537
- [Background] Cole J, Costafreda SG, McGuffin P, Fu CH. Hippocampal atrophy in first episode depression: a meta-analysis of magnetic resonance imaging studies. J Affect Disord. 2011 Nov;134(1-3):483-7. doi: 10.1016/j.jad.2011.05.057. Epub 2011 Jul 13. PMID 21745692
- [Background] Perez-de la Cruz S. Comparison between Three Therapeutic Options for the Treatment of Balance and Gait in Stroke: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jan 7;18(2):426. doi: 10.3390/ijerph18020426. PMID 33430476
- [Background] Cunningham G, Charbonnier C, Ladermann A, Chague S, Sonnabend DH. Shoulder Motion Analysis During Codman Pendulum Exercises. Arthrosc Sports Med Rehabil. 2020 Jun 26;2(4):e333-e339. doi: 10.1016/j.asmr.2020.04.013. eCollection 2020 Aug. PMID 32875297
- [Background] Gribble PA, Kelly SE, Refshauge KM, Hiller CE. Interrater reliability of the star excursion balance test. J Athl Train. 2013 Sep-Oct;48(5):621-6. doi: 10.4085/1062-6050-48.3.03. Epub 2013 Mar 19. PMID 24067151
- [Background] Gujral S, Aizenstein H, Reynolds CF 3rd, Butters MA, Erickson KI. Exercise effects on depression: Possible neural mechanisms. Gen Hosp Psychiatry. 2017 Nov;49:2-10. doi: 10.1016/j.genhosppsych.2017.04.012. PMID 29122145
- [Background] Kubo K, Ikebukuro T, Yata H. Effects of squat training with different depths on lower limb muscle volumes. Eur J Appl Physiol. 2019 Sep;119(9):1933-1942. doi: 10.1007/s00421-019-04181-y. Epub 2019 Jun 22. PMID 31230110
- [Background] Mu L, Cai J, Gu B, Yu L, Li C, Liu QS, Zhao L. Treadmill Exercise Prevents Decline in Spatial Learning and Memory in 3xTg-AD Mice through Enhancement of Structural Synaptic Plasticity of the Hippocampus and Prefrontal Cortex. Cells. 2022 Jan 12;11(2):244. doi: 10.3390/cells11020244. PMID 35053360
- [Background] Pizzagalli DA, Roberts AC. Prefrontal cortex and depression. Neuropsychopharmacology. 2022 Jan;47(1):225-246. doi: 10.1038/s41386-021-01101-7. Epub 2021 Aug 2. PMID 34341498
- [Background] Rottensteiner M, Leskinen T, Niskanen E, Aaltonen S, Mutikainen S, Wikgren J, Heikkila K, Kovanen V, Kainulainen H, Kaprio J, Tarkka IM, Kujala UM. Physical activity, fitness, glucose homeostasis, and brain morphology in twins. Med Sci Sports Exerc. 2015 Mar;47(3):509-18. doi: 10.1249/MSS.0000000000000437. PMID 25003773
- [Background] Shaffer SW, Teyhen DS, Lorenson CL, Warren RL, Koreerat CM, Straseske CA, Childs JD. Y-balance test: a reliability study involving multiple raters. Mil Med. 2013 Nov;178(11):1264-70. doi: 10.7205/MILMED-D-13-00222. PMID 24183777
- [Background] Swift DL, McGee JE, Earnest CP, Carlisle E, Nygard M, Johannsen NM. The Effects of Exercise and Physical Activity on Weight Loss and Maintenance. Prog Cardiovasc Dis. 2018 Jul-Aug;61(2):206-213. doi: 10.1016/j.pcad.2018.07.014. Epub 2018 Jul 9. PMID 30003901
- [Background] Zhang Y, Yang Y, Zhu L, Zhu Q, Jia Y, Zhang L, Peng Q, Wang J, Liu J, Fan W, Wang J. Volumetric Deficit Within the Fronto-Limbic-Striatal Circuit in First-Episode Drug Naive Patients With Major Depression Disorder. Front Psychiatry. 2021 Jan 20;11:600583. doi: 10.3389/fpsyt.2020.600583. eCollection 2020. PMID 33551870